CLINICAL TRIAL: NCT05060848
Title: Plasma Hydrogen Sulfide as a Biomarker for Alzheimer's Disease and Related Dementias
Status: Active, not recruiting | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Elizabeth Ann Disbrow, PhD, Professor, Dept. of Neurology, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: 00000059
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: biomarker; vascular disease; sex differences; race differences
MeSH Terms: conditions — Alzheimer Disease; Dementia; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADRD: Participants in the ADRD group will have a score of greater than or equal to 17 on the ADAS-cog, a paper and pencil test of cognitive function including memory.
  Subgroups based on sex and race categories will also be examined.
- Control: Participants in the control group will have a score of less than 17 on the ADAS-cog, a paper and pencil test of cognitive function including memory

SUMMARY:
Hydrogen sulfide is a signaling molecule that is important for vascular health. Because vascular factors such as hypertension and high cholesterol are risk factors for Alzheimer's disease and related dementias, we hypothesize that hydrogen sulfide plays an important role in brain health as well. We will compare blood levels of hydrogen sulfide across groups of people with and without dementia. We will also look at the relationship between hydrogen sulfide, cognitive dysfunction and measures of brain microvascular disease examine the contribution of hydrogen sulfide to cognitive decline. Our goal is to identify a biomarker of vascular dysfunction in dementia.

DETAILED DESCRIPTION:
We have described hydrogen sulfide (H2S), a signaling molecule important in vascular homeostasis, as a biomarker of cardiovascular disease. There is accumulating evidence that vascular factors such as hypertension, hypercholesterolemia, and type 2 diabetes are associated with increased risk of Alzheimer's disease and related dementias (ADRD). Furthermore, in the brain, H2S acts as a neurotransmitter/second messenger produced following nerve excitation. It also modulates N-methyl-D-aspartate (NMDA) receptors during long term potentiation for memory consolidation. Three biochemical forms of reactive sulfur pools exist: free H2S, acid-labile (e.g. iron-sulfur clusters) and bound sulfide (e.g. persulfides, polysulfides). We hypothesize that H2S becomes dysregulated in ADRD, where vascular and cognitive functions are linked. We will use analytical biochemical methods to measure plasma H2S and its metabolites, and 3T MRI to evaluate indicators of microvascular disease in ADRD. We will compare H2S levels in people with and without cognitive dysfunction consistent with ADRD, and determine the specificity and sensitivity of H2S indistinguishing people with and without cognitive dysfunction. In addition, because previous studies report differences in the incidence and prevalence of ADRD by race and sex, we will compare outcomes across these groups as well. Finally, we will examine the potentially mediating role of H2S in the relationship between cognitive function and microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be aged >55 years with English as the 1⁰ language, with stable permitted medications for <4 weeks, geriatric depression scale score <6, visual and auditory acuity adequate to perform tests, and history of education excluding developmental cognitive abnormalities.

Exclusion Criteria:

* Exclusion criteria are history of significant neurologic disease or mental illness, unstable medical conditions that could interfere with completion of study, substance abuse within 2 years, contraindications to MRI, abnormal findings on MRI, history of chronic kidney disease, and investigational agents within 1 month of participation.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 people with a study based diagnosis of AD (ADAS-cog score ≥17) and 50 controls will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive Outcomes | Prospective, single measurement
  ADAS Cog score
Imaging Outcomes | Prospective, single measurement
  MRI based brain volume measures, FLAIR lesion volume
Blood Outcomes | Prospective, single measurement
  Plasma Hydrogen sulfide including metabolites: free, acid labile, bound and total sulfides.

SECONDARY OUTCOMES:
Demographic Data | Prospective, single measurement
  Age, Race, Sex, Socioeconomic status

OTHER OUTCOMES:
Comorbidity Data (covariates) | Prospective, single measurement
  BP, weight, Hx of smoking, diabetes, hypertension, elevated cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health Shreveport Center for Brain Health, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Disbrow E, Stokes KY, Ledbetter C, Patterson J, Kelley R, Pardue S, Reekes T, Larmeu L, Batra V, Yuan S, Cvek U, Trutschl M, Kilgore P, Alexander JS, Kevil CG. Plasma hydrogen sulfide: A biomarker of Alzheimer's disease and related dementias. Alzheimers Dement. 2021 Aug;17(8):1391-1402. doi: 10.1002/alz.12305. Epub 2021 Mar 12. PMID 33710769